CLINICAL TRIAL: NCT01008228
Title: Comparison of Efficacity of Simple Aspiration Versus Standard Drainage in the Management of Large Size Primary Spontaneous Pneumothorax
Brief Title: Comparison of Exsufflation Versus Drainage in Primary Spontaneous Pneumothorax
Acronym: EXPRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Belfort Hospital (Other); Central Hospital, Nancy, France (Other); Norman Bethune Medical Hospital (Other); St Philibert Hospital, Lomme (Unknown); Hospital of Montfermeil (Unknown); University Hospital, Brest (Other); University Hospital, Clermont-Ferrand (Other); Nantes University Hospital (Other); Association Hospitalière Nord Artois Cliniques (Other); Poitiers University Hospital (Other); University Hospital, Tours (Other); CHU de Reims (Other); Centre hospitalier de Perpignan (Other); Hospices Civils de Lyon (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Hospital of Roubaix (Unknown); Hospital of Boulogne/mer (Unknown); Assistance Publique Hopitaux De Marseille (Other); University Hospital, Rouen (Other); University Hospital, Angers (Other Government); Centre Hospitalier le Mans (Other); Centre Hospitalier Universitaire de Nīmes (Other); University Hospital, Grenoble (Other); Hospital of Mulhouse (Unknown); Hospital of Valence (Unknown)
Responsible Party: Principal Investigator, DESMETTRE, Dr Thibaut Desmettre, MD, PhD, Centre Hospitalier Universitaire de Besancon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R/2009/38
Record Dates: First submitted 2009-09-09; First posted 2009-11-05 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Pneumothorax
Keywords: spontaneous; primary; first episode
MeSH Terms: conditions — Pneumothorax | interventions — Chest Tubes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tube thoracic drainage (Active Comparator): drainage performed with tube drainage CH 16 or ch 20
  Interventions: Procedure: thoracic tube drainage
- exsufflation (Experimental): exsufflation with a specific thoracentesis system
  Interventions: Procedure: exsufflation

INTERVENTIONS:
Procedure: exsufflation — exsufflation will be performed with a specific thoracentesis system after introducing the device into chest pneumothorax, aspiration will be performed during 30 minutes
  Other Names: Turkel Kit
  Arms: exsufflation
Procedure: thoracic tube drainage — thoracic tube drainage will be performed with a tube Ch 16 or ch 20
  Other Names: Monod Trocar; Chest Tube
  Arms: tube thoracic drainage

SUMMARY:
Management of primary spontaneous pneumothorax (PSP) remains unclear. Primary therapeutic goals for PSP include removal of air from the pleural space an prevention of recurrences. The absence of generally accepted and methodologically sound recommendations may account for the extensive variation in practice for air evacuation techniques. Air evacuation may be achieved by simple aspiration (exsufflation) or conventional chest tube drainage. Chest tube thoracotomy remains the most popular technique.Aspiration is a more simple technique, that allows possibility of ambulatory management. The purpose of the present study is to compare simple aspiration performed with a specific thoracentesis device, versus conventional chest tube drainage. Comparison will be performed on immediate efficacity of resolution of the pneumothorax.The hypothesis is that simple aspiration performed with a specific device is not inferior to chest tube drainage for management of a first episode of large size primary spontaneous pneumothorax. A second goal is to measure the efficacy at one week, and the recidive at one year. The trial is randomized, controlled and will include 200 patients for each group. The patients will be enrolled in 29 hospitals in France. Emergency department, thoracic surgery and pulmonary departments of each hospital were primarily contacted for agreement to participate to the study.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 18 years and less than 50 years
* first episode of pneumothorax
* primary pneumothorax (absence of known pulmonary disease)
* large size of pneumothorax : presence of a visible rim of air between the lund margin and the chest wall, from the apex to pulmonary base

Exclusion Criteria:

* impossibility to obtain patient consent for psychiatric disease
* patients under justice control
* âgé less than 18 years, or more than 50 years
* impossibility of medical follow de for geographic, social or psychic reasons
* pregnant women
* pneumothorax with acute respiratory insufficiency or bad tolerated
* recidive of pneumothorax
* traumatic pneumothorax
* pneumothorax with pleural effusion
* bilatéral pneumothorax
* pneumothorax with pulmonary disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 402 (Actual)
Dates: Start 2009-06; Primary Completion 2014-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
size of residual pneumothorax measured on chest radiography | one day

SECONDARY OUTCOMES:
size of residual pneumothorax at one week | one week
recidive of pneumothorax at one year | one year

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut TJ Desmettre, Principal Investigator — Hospital University of Besancon; Thibaut DESMETTRE, MD, Principal Investigator — CHU Besançon
Locations (24):
- France (24):
  - Centre Hospitalier Intercommunal de la Haute Saône, Vesoul, Franche Comté
  - CHU Angers, Angers
  - Hôpital Henri Mondor, Aurillac
  - Centre Hospitalier, Belfort
  - CHU Besancon, Besançon
  - CH Bethune, Béthune
  - CH Boulogne sur Mer, Boulogne-sur-Mer
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Clinique de HENIN BEAUMONT, Hénin-Beaumont
  - CH Lomme, Lomme
  - CHU Marseille, Marseille
  - Chi Le Raincy/Montfermeil, Montfermeil
  - CH Mulhouse, Mulhouse
  - CHU Nimes, Nîmes
  - CH Perpignan, Perpignan
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHR Roubaix, Roubaix
  - CH Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Background] Desmettre T, Meurice JC, Kepka S, Dalphin JC. [Treatment of first spontaneous pneumothorax: drainage or exsufflation?]. Rev Mal Respir. 2011 Jan;28(1):5-8. doi: 10.1016/j.rmr.2010.10.028. Epub 2011 Jan 12. No abstract available. French. PMID 21277468
- [Background] Desmettre T, Meurice JC, Mauny F, Woronoff MC, Tiffet O, Schmidt J, Ferretti G, Dalphin JC. [Comparison of simple aspiration versus standard drainage in the treatment of large primary spontaneous pneumothorax]. Rev Mal Respir. 2011 Mar;28(3):336-43. doi: 10.1016/j.rmr.2010.10.030. Epub 2011 Mar 10. French. PMID 21482337
- [Background] Desmettre T, Meurice JC, Tapponnier R, Pretalli JB, Dalphin JC. [The EXPRED study: where are we?]. Rev Mal Respir. 2013 Jan;30(1):18-21. doi: 10.1016/j.rmr.2012.09.019. Epub 2012 Nov 13. No abstract available. French. PMID 23318185
- [Derived] Marx T, Joly LM, Parmentier AL, Pretalli JB, Puyraveau M, Meurice JC, Schmidt J, Tiffet O, Ferretti G, Lauque D, Honnart D, Al Freijat F, Dubart AE, Grandpierre RG, Viallon A, Perdu D, Roy PM, El Cadi T, Bronet N, Duncan G, Cardot G, Lestavel P, Mauny F, Desmettre T. Simple Aspiration versus Drainage for Complete Pneumothorax: A Randomized Noninferiority Trial. Am J Respir Crit Care Med. 2023 Jun 1;207(11):1475-1485. doi: 10.1164/rccm.202110-2409OC. PMID 36693146